CLINICAL TRIAL: NCT03628846
Title: A Prospective Survey of Opioid Use After Traumatic Injury in Adolescents
Brief Title: Opioid Use After Traumatic Injury in Adolescents
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Olena Mazurenko, Associate Professor of Health Policy, Indiana University
Other Study IDs: 1706176501
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Opioid Use; Traumatic Injury; Adolescent Behavior; Substance Abuse Disorder
MeSH Terms: conditions — Wounds and Injuries; Adolescent Behavior; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva will be collected at baseline only for the purpose of analyzing genetic data on each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traumatically Injured Adolescent
- Not Traumatically Injured Adolescent

SUMMARY:
Currently, 1 in 8 adolescents continue to receive prescription opioids a year or more after injury. By longitudinally surveying patients, we can identify risk factors and pathways to nonmedical opioid use. Furthermore, by assessing whether pain management and mental health treatment after injury moderates sustained opioid use and prescription opioid misuse, we can create targeted interventions to reduce future nonmedical opioid use in adolescents.

DETAILED DESCRIPTION:
This is a prospective cohort study that will follow participants for 2 years and administer surveys to adolescents both traumatically injured and uninjured on prescription opioid usage, substance use, utilization of pain management and mental health services, and mental and physical health condition conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 12-20 years of age
* Adolescent admitted for trauma OR adolescent with no recent trauma
* English speaking
* Consent can be obtained from a parent or guardian

Exclusion Criteria:

- Patients with severe brain injuries or other injuries that prevent survey participation

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Traumatically injured patients admitted to either Eskenazi Hospital or Riley Hospital, between the ages of 12 and 20.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Prospectively determine drivers of sustained opioid use and prescription opioid misuse. | 2 years

SECONDARY OUTCOMES:
Identify patient-reported factors for sustained prescription opioid use, including chronic pain and mental health conditions such as PTSD, depression, anxiety, and sleep disorders. | 2 years
Assess behavioral, social, and clinical predictors of prescription opioid misuse and nonmedical opioid use by longitudinally surveying injured adolescents. | 2 years
Qualitatively determine patients' motives for continued opioid therapy, prescription opioid misuse, and nonmedical opioid use by interviewing injured adolescents. | 2 years
Analyze genetic information, obtained via saliva sample and the company 23andMe, from each participant to determine if some people are more likely to use more pain medication than others or respond better to certain pain medications. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided